CLINICAL TRIAL: NCT00651365
Title: A Phase I Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of the Selective Met Inhibitor JNJ-38877605 in Subjects With Advanced or Refractory Solid Tumors
Brief Title: A Safety and Dose-finding Study of JNJ-38877605 in Patients With Advanced or Refractory Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early termination due to increase in serum creatinine levels and minimal PD activity.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Director, Clinical Scientist, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014644; CR014644 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Neoplasms
Keywords: Advanced solid tumors; Refractory solid tumor; Antineoplastic protocol; Drug therapy; Pharmacokinetics; Met inhibitor
MeSH Terms: conditions — Neoplasms | interventions — JNJ38877605

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 001 (Experimental)
  Interventions: Drug: JNJ-38877605

INTERVENTIONS:
Drug: JNJ-38877605

SUMMARY:
This purpose of the study is to determine what dose of JNJ-38877605 is safe and if JNJ-38877605 has any effect in patients with advanced or refractory solid tumors for which there are not alternative therapies.

DETAILED DESCRIPTION:
JNJ-38877605 is a new drug being developed for the treatment of cancer. It is an inhibitor of mesenchymal epithelial transition (Met) kinase, a substance identified in many cancers. This is the first study in which JNJ-38877605 will be administered in man. This research study is being carried out to determine the highest dose of JNJ-38877605 that patients with advanced or refractory solid tumors can tolerate. The study will also test the safety of JNJ-38877605. Safety evaluations will include an assessment of adverse events, clinical laboratory data, electrocardiograms, vital signs measurements, physical examination findings, and Eastern Oncology Cooperative Group (ECOG) performance status. In some patients the effect of food on how the drug is absorbed will also be studied. Throughout the study, treatment will be given in cycles which will be 21 days long and the study drug will be taken once a day. The number of cycles will depend on the effects the drug has on the patient and whether the patient benefits from the treatment. The design of a cycle may be adjusted during the course of the study, so that the cycle is shorter or longer, or includes some days when the patient does not receive treatment (a pause = intermittent treatment). It is also possible the drug will be taken more than once a day. In case of any changes to the drug administration schedule, the schedule and the timing of visits and blood/urine tests may be adapted accordingly, without increasing their number. During the first treatment cycle, 2 or 3 overnight stays in the hospital are required and visits to the hospital during cycles 1, 2, 3, and 4 may take up to 12 hours after the morning dose. From cycle 5 onwards, there is a daytime visit only once every cycle, and these usually take up less time. Patients are informed about the current visit schedule at enrollment and throughout the study. The dose of JNJ-38877605 administered in the study will start low and will be increased during the study. The amount of study drug taken each day by an individual patient depends on when the patient enrolls in the study. If a group of patients does not have severe side effects, the next group of patients will get a higher dose. The dose will increase until some patients have severe side effects. The dose will then be decreased and 3 to 6 patients will receive the highest amount of drug where severe side effects were not observed. The amount of JNJ-38877605 in the patient's blood will be measured and the study will also look at the effect of the drug on the disease. The patient may continue treatment as long as there is benefit as assessed by the response assessments throughout the study and the patient has no unacceptable side effects. A follow-up visit for each patient will take place within 14 days after the patient takes the last dose of JNJ-38877605. JNJ-38877605 is provided in 10, 50, and 100 mg capsules for oral use. JNJ-38877605 will initially be administered once a day orally although the administration schedule may be modified at later stages in the study. JNJ-38877605 will be provided as a take-home formulation in childproof high-density polyethylene bottles.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced or refractory solid tumor no longer eligible for approved therapies
* Eastern Cooperative Oncology Group performance status test score of <=2
* Must meet protocol lab criteria which will include lab assessment of adequate bone marrow function, liver function, and renal function.

Exclusion Criteria:

* Any medical condition that requires wound healing during the study (for example chronic leg ulcers, gastric ulcer disease, or expected major surgery)
* Major surgery within 3 weeks before enrollment
* Decreased or deficient coagulability of blood (for example genetic defects such as protein Z deficiency) or compliance problems in subjects required to take anticoagulants (e.g., coumarin derivates, acetylsalicylic acid) which could result in decreased or deficient coagulability
* Chemotherapy (for nitrosoureas and mitomycin C within 6 weeks), radiotherapy, immunotherapy, or any other investigational agent within 3 weeks before study drug administration
* antibody therapy within 3 months before administration of JNJ-38877605
* brain metastases
* History of uncontrolled heart disease within 12 months before enrollment or any protocol-defined cardiovascular abnormalities
* Patients with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of JNJ-38877605 by assessment of the adverse event profile (throughout the study), dose-limiting toxicity (Cycle 1), and the maximum tolerated dose.

SECONDARY OUTCOMES:
Determine the pharmacokinetic profile of JNJ-38877605 and its metabolite, JNJ-40434654 and to investigate the potential impact of food on the PK profile (Cycle 1). Explore the pharmacodynamic effects and measure anti-tumor activity of JNJ-38877605.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.